CLINICAL TRIAL: NCT00613197
Title: A One Year, Multi-center, Randomised, Double-blind Placebo-controlled Parallel-groups Assessment of the Tolerability, Safety and Efficacy of Epanova Soft Gelatin Capsules 4g/Day for Maintenance of Remission of Crohn's Disease.
Brief Title: EPANOVA in Crohn's Disease, Study 1
Acronym: EPIC-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Prof. P. Rutgeerts, University of Leuven, Belgium
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP0307
Record Dates: First submitted 2008-01-15; First posted 2008-02-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Epanova (Experimental)
  Interventions: Drug: Epanova
- 2 Placebo (Placebo Comparator)
  Interventions: Drug: Epanova

INTERVENTIONS:
Drug: Epanova — 4g/day in divided doses

SUMMARY:
The primary objective of this study is to assess the ability of EpanovaTM Soft Gelatin Capsules at a total daily dose of 4g (4x 1g capsules) to maintain remission (Crohn's Disease Activity Index CDAI < 150) in CD patients in whom remission, stable for at least three months and no longer than one year, has been induced by corticosteroids, azathioprine/6-MP, methotrexate, 5-ASA or antibiotics.

Secondary objectives are to assess the:

efficacy of Epanova versus placebo by Crohn's Disease Activity Index (CDAI), Investigator and Subject Global Ratings, employment status and use of CD related medical visits in subjects with CD in remission

safety and tolerability of Epanova

ability of Epanova to maintain the quality of life of CD patients in remission

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, age 17 or older; country-specific age limitations will be followed
2. Diagnosis of Crohn's disease confirmed by radiological studies or endoscopy or surgical pathology within 36 months prior to randomisation
3. In remission for at least 3 months, but no longer than 12 months; remission being defined as meeting both of the two conditions: (1) clinically in remission with a CDAI of less than 150 and (2) off steroids and/or immunosuppressants for at least 3 months, if remission had been induced with such medications

Exclusion Criteria:

1. Intolerance of omega-3 fatty acids or known allergy to fish or fish products
2. Ongoing CD therapy with: 5-ASA compounds, steroids, immune modifiers, systemic antibiotics, tube feeding, defined formula diets or parenteral nutrition
3. In 3 months prior to randomisation received: systemic steroid therapy, azathioprine, 6-mercaptopurine, methotrexate, cyclosporine, probiotic products or preparations containing fish oil
4. In 12 months prior to randomisation received: biologicals e.g. enbrel, infliximab, mycophenolate, tacrolimus, thalidomide, other immune modifiers and/or investigational products
5. Chronic use of narcotics for pain control (opiates for diarrhoea are acceptable)
6. Documented short bowel syndrome, ostomy
7. Need for bowel surgery for CD, bowel obstruction or resection in past 3 months (a subject who had a bowel resection in the past must have had at least one relapse after the surgery)
8. Malignancy and/or clinically significant impairment in cardiac, liver or renal function, CNS, pulmonary, hematological, immunological, vascular and gastrointestinal disease in addition to CD
9. Known alcoholism or drug abuse
10. Any medical conditions which, in the investigator's opinion, may interfere with the evaluation of the trial medication
11. Any of the following laboratory abnormalities:

    * White blood count < 3 x 109/L
    * Lymphocyte count < 0.5 x 109/L
    * Haemoglobin < 80 g/L
    * Platelet count < 125 x 109/L or > 800 x 109/L
    * ALT or AST > 2.0 times the upper limit of normal
    * Alkaline Phosphatase > 2.0 times the upper limit of normal
    * Serum Creatinine > 1.5 times the upper limit of normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2003-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
time to clinical relapse | 52 weeks

SECONDARY OUTCOMES:
CDAI Investigator and subject global rating Quality of life C-reactive protein | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rutgeerts, MD, Prof., Principal Investigator — University of Leuven
Locations (1):
- University of Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Feagan BG, Sandborn WJ, Mittmann U, Bar-Meir S, D'Haens G, Bradette M, Cohen A, Dallaire C, Ponich TP, McDonald JW, Hebuterne X, Pare P, Klvana P, Niv Y, Ardizzone S, Alexeeva O, Rostom A, Kiudelis G, Spleiss J, Gilgen D, Vandervoort MK, Wong CJ, Zou GY, Donner A, Rutgeerts P. Omega-3 free fatty acids for the maintenance of remission in Crohn disease: the EPIC Randomized Controlled Trials. JAMA. 2008 Apr 9;299(14):1690-7. doi: 10.1001/jama.299.14.1690. PMID 18398081